CLINICAL TRIAL: NCT03407105
Title: A Phase I, Open-Label, Dose-Escalation Study of MDX-010 Administered Monthly as Immunotherapy in Subjects Infected With Human Immunodeficiency Virus
Brief Title: A Dose-Escalation Study of MDX-010 Administered Monthly as Immunotherapy in Subjects Infected With Human Immunodeficiency Virus (HIV)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Medarex (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDX010-10
Record Dates: First submitted 2018-01-17; First posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Human Immunodeficiency Virus (HIV)
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 2 (Experimental): Specified dose on specified days
  Interventions: Biological: MDX-010

INTERVENTIONS:
Biological: MDX-010 — Specified dose on specified days
  Other Names: Ipilimumab; BMS-734016

SUMMARY:
The purpose of this study is to assess the safety and tolerability of 2 or 4 doses of MDX-010 in HIV-infected subjects

ELIGIBILITY:
Inclusion Criteria:

* Detectable HIV viremia (HIV-1 RNA level between 1,000 and 100,000 copies/mL)
* CD4 count greater than or equal to 100 cells/mm3
* Current antiretroviral therapy regimen following at least 2 previous changes for documented virologic failure
* Documented resistance tests demonstrating the presence of at least 1 mutation to each major therapeutic class of antiretroviral therapy
* No significant organ compromise

Exclusion Criteria:

* Initiation of any new medications that might reasonably affect the immune response or viral load within 4 weeks prior to screening
* Tetanus booster immunization within 2 months of screening, or a history of anaphylaxis or severe local reaction to the tetanus vaccine
* History of autoimmune disease at risk for recurrence
* Current malignancy, except Stage A or B cervical carcinoma or basal cell carcinoma
* Chronic viral hepatitis, due to Hepatitis B or Hepatitis C undergoing current treatment or Hepatitis B DNA greater than 25 pg/cc or Hepatitis C RNA greater than 20,000 IU/cc
* Currently undergoing treatment or prophylaxis for tuberculosis infection
* Chronic active infectious disease (other than HIV)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 24 (Actual)
Dates: Start 2003-04-21 (Actual); Primary Completion 2006-02-21 (Actual); Study Completion 2006-02-21 (Actual)

PRIMARY OUTCOMES:
Number of treatment induced dose limiting toxicities (DLTs) | Up to 141 days
Grade of treatment induced DLTs | Up to 141 days
Number of treatment emergent AEs (adverse events) | Up to 141 days

SECONDARY OUTCOMES:
Maximum plasma concentration observed post-dose (Cmax) | Up to 141 days
Time of maximum plasma concentration observed post-dose (Tmax) | Up to 141 days
HIV Ribonucleic Acid (RNA) level | Up to 141 days
CD4 (cluster of differentiation) T (thymus) cell cytokine responses to Human Immunodeficiency Virus-1 (HIV-1) antigens | Up to 141 days
CD4 T cell cytokine responses to Candida antigen | Up to 141 days
CD4 T cell cytokine responses to tetanus antigen | Up to 141 days
CD8 (cluster of differentiation) T cell cytokine responses to HIV-1 antigens | Up to 141 days
CD8 T cell cytokine responses to Candida antigen | Up to 141 days
CD8 T cell cytokine responses to tetanus antigen | Up to 141 days
Lymphocyte Proliferation Assay (LPA) to HIV-1 antigens | Up to 141 days
LPA to Candida antigens | Up to 141 days
LPA to tetanus antigens | Up to 141 days
Anti-tetanus toxin antibody level | Up to 141 days
Number of CD4 T cells | Up to 141 days
Number of CD8 T cells | Up to 141 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (5):
- United States (5):
  - Tower ID Medical Associates, Los Angeles, California
  - Quest Clinical Research, San Francisco, California
  - Care Resource, Miami, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Shannon Schrader, MD, Houston, Texas

REFERENCES:
- [Derived] Colston E, Grasela D, Gardiner D, Bucy RP, Vakkalagadda B, Korman AJ, Lowy I. An open-label, multiple ascending dose study of the anti-CTLA-4 antibody ipilimumab in viremic HIV patients. PLoS One. 2018 Jun 7;13(6):e0198158. doi: 10.1371/journal.pone.0198158. eCollection 2018. PMID 29879143